CLINICAL TRIAL: NCT04375449
Title: Investigation of Milk Peptides (Pep2Dia®) on Postprandial Blood Glucose Profile in Prediabetic Subjects: Randomized, Double-blind, Placebo-controlled, Cross-over Study With Different Dosages
Brief Title: Investigation of Milk Peptides (Pep2Dia®) on Postprandial Blood Glucose Profile in Prediabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredia S.A. (Industry)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTS1472/20
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: The study will be performed as a multicentric, randomized, double-blind, and placebo-controlled in a 3-way cross-over design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pep2dia- dosage 1 (Active Comparator): 700mg of whey protein hydrolysates single dose
  Interventions: Dietary Supplement: Pep2dia
- Pep2Dia - dosage 2 (Active Comparator): 1400mg of whey protein hydrolysates single dose
  Interventions: Dietary Supplement: Pep2dia
- Placebo (Placebo Comparator): maltodextrin single dose
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Pep2dia — what is the effect of Pep2dia on postprandial glycemia after a meal rich in carbohydrates (75g)
  Arms: Pep2Dia - dosage 2; Pep2dia- dosage 1
Dietary Supplement: maltodextrin — maltodextrin
  Arms: Placebo

SUMMARY:
The goal is to investigate the 180 min postprandial response on blood glucose and insulin levels after intake of Pep2Dia® in two different dosages compared to placebo in the context of a meal challenge test, providing 75 g of carbohydrates. Pep2Dia® will be administered 15 min prior to a standardized challenge meal.

DETAILED DESCRIPTION:
From a previous pilot study (BTS1130/17) there is first evidence that the native whey product with alpha-glucosidase inhibiting properties (Pep2Dia®) has the potential to modulate postprandial hyperglycaemia in prediabetic subjects.

Thereby, incremental areas under the curve (iAUC) of glucose as the primary outcome were significantly reduced by a single dosage of 1400 mg Pep2Dia® compared to placebo the second study is to investigate the 180 min postprandial response on blood glucose and insulin levels after intake of Pep2Dia® in two different dosages compared to placebo in the context of a meal challenge test, providing 75 g of carbohydrates. Pep2Dia® will be administered 15 min prior to a standardized challenge meal. Furthermore, the 120 min postprandial incretin response in terms of Glucagon-like Peptide-1 (GLP-1) will be determined. Changes in insulin sensitivity will be determined by the Matsuda-index as appropriate outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects (minimum one third of each gender) with prediabetic HbA1c values between 5.7% - 6.4% and/or fasting glucose ≥ 5.6 mmol/L (≥ 100 mg/dL) and < 7.0 mmol/L (< 125 mg/dL) (in venous plasma) (twice confirmed at two independent days if HbA1c is < 5.7%)
* Body mass index 19-35 kg/m2
* Non-smoker
* Caucasian
* Availability and presence in the study units for approx. 3.5 hours/ week for 3 times.
* Signed informed consent form
* No changes in food habits or physical activity 3 months prior to screening and during the study

Exclusion Criteria:

* Presence of disease or drug(s) influencing digestion and absorption of nutrients or bowel habits
* Intake of medications known to affect glucose tolerance, e.g., diabetic medication, steroids, protease inhibitors or antipsychotics
* Diagnosed Typ 2-Diabetics with medical treatment
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid (100 mg as standard prophylactic treatment allowed when dose is stable 1 month prior to screening), anticoagulants, diuretics, thiazides (diuretics and thiazides allowed e.g. for hypertension treatment when dose is stable 1 month prior to screening)), which in the Investigator's opinion would impact patient safety
* Severe liver, renal or cardiac disease
* Acute gastrointestinal diseases including diarrhea and/or vomiting within the last 2 weeks
* Known inflammatory and malignant gastrointestinal diseases (i.e. colitis ulcerosa, Morbus Crohn, celiac disease, malignant diseases e.g. colon-cancer, rectum cancer, pancreatitis)
* Clinically relevant findings as established by medical history, physical examination, clinical laboratory and/or vital signs
* Major medical or surgical event requiring hospitalization within the previous 3 months
* Intake of antibiotics within 4 weeks before the test days
* Known alcohol abuse or drug abuse
* Pregnant or breast feeding women
* Known or suspected allergy to any component of the investigational product(s) (e.g. milk protein)
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study
* Subject unable to co-operate adequately

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Glucose-iAUC(0-180min) | Day 1, Day 15, Day 29
  Area under the curve calculated as the incremental area under the blood glucose response curve, ignoring the area beneath the fasting concentration (according to ISO 26642:2010(E)

SECONDARY OUTCOMES:
Cmax | Day 1, Day 15, Day 29
  Maximum blood glucose concentration
Max_increase | Day 1, Day 15, Day 29
  Cmax minus baseline value
Tmax | Day 1, Day 15, Day 29
  Time to reach maximum blood glucose concentration
Tbaseline | Day 1, Day 15, Day 29
  First time to reach baseline again after increase or decrease in blood glucose
AUC(0-180min) | Day 1, Day 15, Day 29
  Total area under curve from 0 to 180 min for blood glucose concentration
Matsuda index | Day 1, Day 15, Day 29
  Marker of insulin sensitivity
Increase of insulin | Day 1, Day 15, Day 29
  Area under the curve calculated as the incremental area under the Insulin response curve, ignoring the area beneath the fasting concentration (Insulin-iAUC(0-180min)). If applicable further pharmacokinetic data from insulin increase will be calculated (e.g. Cmax, Tmax)
GLP-1-iAUC(0-120min) | Day 1, Day 15, Day 29
  120 min postprandial incretin response in terms of Glucagon-like Peptide-1

CONTACTS AND LOCATIONS:
Locations (1):
- Biotesys, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No